CLINICAL TRIAL: NCT03519841
Title: Performance Study of a Non-invasive Glucose Monitoring Device Prototype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: RSP-13
Record Dates: First submitted 2018-04-11; First posted 2018-05-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Non-randomized interventional study comparing device and blood reference measurements in diabetic patients
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSP-13-01 (Experimental): Experimental: IMD data collection Subjects will intensively collect spectral Raman data on P0.1 in a home-based setting for 5 days. Data will be paired with reference measurements.
  Interventions: Device: P0.1
- RSP-13-02 (Experimental): Experimental: IMD data collection Subjects will collect spectral Raman data on P0.1 during four measuring sessions a day for 30 days distributed over a time period of 60 days. Each timepoint is conducted in duplicate. Spectral data will be compared to standard BG measurements.
  Interventions: Device: P0.1

INTERVENTIONS:
Device: P0.1 — Investigational Medical Device collecting spectral Raman data from tissue.

SUMMARY:
This clinical study has been launched to collect spectral Raman data paired with validated glucose reference values in private homes of subjects.

DETAILED DESCRIPTION:
Protocol consists of two parts:

Part A) Subjects will collect spectral Raman data on device every 15 minutes for 10 hours a day for five days. The five days will be distributed within a timeframe of ten days. A Flash Glucose Monitor will be used as a comparator. In addition to this, four daily capillary Blood Glucose readings will be collected.

Part B) Subjects will perform four daily measuring sessions in which optical Raman readings are paired with capillary Blood Glucose comparator. Measuring sessions are performed in subjects' own home while maintaining usual diabetes management routines. Subjects will collect data for 30 days during a 60 days' period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older
* Diabetic patients (all types), insulin requiring
* Skin phototype 1-4

Exclusion Criteria:

* For female participants: Pregnancy or subject is attempting to conceive or not willing and able to practice birth control during the study duration
* For female participants: Breastfeeding
* Subjects not able to understand and read Danish
* In Investigator's opinion, subject is not able to follow instructions as specified in the protocol
* Rejection by optical screenings
* Participants not able to hold hand/arm steadily (including tremors and Parkinson's Disease)
* Diagnosed with reduced circulation
* Extensive skin changes, tattoos or diseases on probe application site
* Known allergy to medical grade alcohol
* Known allergy to adhesives, applicable to subjects in RSP-13-01
* Systemic or topical administration of glucocorticoids for the past 7 days
* Subjects undergoing dialysis treatment
* Medical history or any condition that may, in the opinion of the Investigator, compromise the subject's ability to participate
* Concomitant medical condition which could present a risk to the safety or welfare of the subject or study staff.
* Participants currently enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Generation and validation of predictive models by ISUP and MARD measures | 6 months
  Optical glucose data will be collected together with paired reference values (BGM and FGM, Protocol 1 and BGM, Subprotocol 2).
  For subprotocol 1, measurements will be collected every 15 minutes for 10 hours a day for 5 days distributed over a period of 10 days.
  For subprotocol 2, four daily measurements will be collected while subject is maintaining normal routines. Data will be collected for 30 days distributed over a period of 60 days.
  Optical glucose readings will be masked to the subjects.
  Collected data will be used to generate individual calibration models capable of predicting tissue glucose. Models will be validated on independent data sets using MARD and ISUP measures.

SECONDARY OUTCOMES:
Safety evaluation: paucity of adverse events | 6 months
  Safety will be evaluated in a descriptive manner by the paucity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Henriksen, MD, PhD, Principal Investigator — Steno Diabetes Center Odense, Denmark; Vibe Vestergaard, Nurse, Principal Investigator — Steno Diabetes Center Odense, Denmark
Locations (1):
- Steno Diabetes Center Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No